CLINICAL TRIAL: NCT05424640
Title: Intervention of Specific Dietary Fibers on Dynamics of Individual Gut Microbiota
Brief Title: Dietary Fiber and Gut Microbiome Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center of Food and Fermentation Technologies (Other)
Responsible Party: Principal Investigator, Kaarel Adamberg, Project manager, Center of Food and Fermentation Technologies
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: RTKU
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Healthy
Keywords: Gut microbiome; food diary; dietary fibers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Baseline (No Intervention): Collection of baseline data 1 week before intervention
- Dietary fiber 1 (Experimental): 15 g/day oat fiber 3 weeks intervention
  At the end of period following analyses are collected:
  1 week food diary blood sample microbiome sample gut health questionnaire
  Interventions: Dietary Supplement: Dietary fiber 1
- Wash-out 1 (No Intervention): 2 weeks
  At the end of period following analyses are collected:
  1 week food diary blood sample microbiome sample gut health questionnaire
- Dietary fiber 2 (Experimental): 15 g/day dietary fiber mix I 3 weeks intervention
  At the end of period following analyses are collected:
  1 week food diary blood sample microbiome sample gut health questionnaire
  Interventions: Dietary Supplement: Dietary fiber 2
- Wash-out 2 (No Intervention): 2 weeks
  At the end of period following analyses are collected:
  1 week food diary blood sample microbiome sample gut health questionnaire
- Dietary fiber 3 (Experimental): 15 g/day dietary fiber 3 3 weeks intervention
  At the end of period following analyses are collected:
  1 week food diary blood sample microbiome sample gut health questionnaire
  Interventions: Dietary Supplement: Dietary fiber 3
- Wash-out 3 (No Intervention): 2 weeks
  At the end of period following analyses are collected:
  1 week food diary blood sample microbiome sample gut health questionnaire
- Dietary fiber 4 (Experimental): 15 g/day rye fiber 3 weeks intervention
  At the end of period following analyses are collected:
  1 week food diary blood sample microbiome sample gut health questionnaire
  Interventions: Dietary Supplement: Dietary fiber 4
- Wash-out 4 (No Intervention): 2 weeks
  At the end of period following analyses are collected:
  1 week food diary blood sample microbiome sample gut health questionnaire

INTERVENTIONS:
Dietary Supplement: Dietary fiber 1 — Description in the arm description
  Arms: Dietary fiber 1
Dietary Supplement: Dietary fiber 2 — Description in the arm description
  Arms: Dietary fiber 2
Dietary Supplement: Dietary fiber 3 — Description in the arm description
  Arms: Dietary fiber 3
Dietary Supplement: Dietary fiber 4 — Description in the arm description
  Arms: Dietary fiber 4

SUMMARY:
The purpose of this dietary intervention is to study the effects of several dietary fibers on the gut microbiota at the personal level. Hypothesis 1: Intake of specific dietary fibers improves the blood lipid profile depending on the personal microbiota of the participants.

Hypothesis 2: detailed food intake analysis and continuous monitoring of gut microbiota enables to draw causative interrelationships between food components, bacteria of gut microbiome and health characteristics.

DETAILED DESCRIPTION:
The study design is a cross-over, pre-post intervention trial. All participants are enrolled into all study periods. Study consists of baseline period, four periods of dietary fiber intervention and four periods of wash-outs.

The main goal of this study was to elucidate the patterns between individual dietary fibers and gut microbiota at the personal level. Each person has a unique (individual) intestinal microbiological profile that changes according to lifestyle (diet, environment, physical activity), age and health status. With next generation sequencing methods to map microbial communities and detailed nutritional analysis including blood tests, it is possible to identify the specific effects of specific fiber on a selected (individual) microbiota. TFTAK researchers have long-term experience in microbiota analysis as well as diet design and nutrition analysis, which can be successfully applied in this project.

PRELIMINARY STUDY EVALUATION AND TESTING

1. Complete preliminary study questionnaire
2. Complete orientation to the study and provide voluntary consent to join the study
3. Collection of coded intervention products, sampling supplies, and instructional materials

1-WEEK QUESTIONNAIRE AND LABORATORY VISIT

1. Record food intake and gastrointestinal function for 7 days 2. Collect health data and provide a 7-day food diary using web-based program Nutridata (tap.nutridata.ee) 3. Provide a stool and blood sample at the laboratory 3-WEEK QUESTIONNAIRE AND

LABORATORY VISITS

1. Record food intake and gastrointestinal symptoms for 7 days
2. Collect health data and provide a 3-day food frequency questionnaire
3. Provide a stool and blood sample at the laboratory BLOOD SAMPLE

ANALYSES

1. Provide the blood sample at the laboratory in the morning in an overnight fasted state.

DIETARY INTERVENTION

Study consists of baseline period, four periods of dietary fiber intervention and four periods of wash-outs:

1. Baseline mapping (health questionnaire, 1 week food diary before sampling of blood and gut microbiota)
2. Dietary fiber 1, 3 weeks, analyses: health questionnaire, 1 week food diary before sampling of blood and gut microbiota
3. Wash-out period, 2 weeks, analyses: health questionnaire, 1 week food diary before sampling of blood and gut microbiota
4. Repeating 3 times periods of 2 and 3. In each dietary fiber period 15 g/day of oat fiber, rye fiber, mix I and mix II of dietary fibers are used as test compounds. Dietary fiber mix I and mix II are inulin, beta-glucan, polydextrose, citrus pectin and psyllium, and beta-glucan, citrus pectin and psyllium, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-60

  * Normal bowel function
  * Omnivorous diet
  * Ability to provide a signed written informed consent
  * Willing to provide stool and blood specimens over the 22-week study period

Exclusion Criteria:

* Diagnosed history of chronic diseases including coronary heart disease, stroke, cancer, type 1 or 2 diabetes mellitus, inflammatory bowel disease, gastritis, autoimmune disease, or rheumatoid arthritis

  * Medication: statins, blood pressure medications, antidepressants, other prescription medications
  * History of bariatric operation, removal of the gallbladder.
  * Food allergies, lactose intolerance
  * Recent (previous 3 months) use of antibiotics
  * Intake of highly dosed pre- or probiotics 2 weeks prior and during the study
  * Current pregnancy or breastfeeding
  * Volunteers showing previously unrecognized illness will also be excluded
  * Individual unable to give informed consent

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of the intestinal microbiota | 150 days
  Fecal microbiota analysis based on the 16S ribosomal RNA (rRNA) sequencing pre- and post-dietary intervention.
Evaluation of food consumption data | 150 days
  All foods consumed were collected 1 week before the end of every study period using web-based program (tap.nutridata.ee)
Evaluation of blood lipid profile | 150 days
  Triglycerides, total cholesterol, HDL-cholesterol, LDL-cholesterol after every intervention and wash-out in plasma (mmol/L).
Evaluation of blood glucose levels | 150
  Fasting glucose pre- and post-dietary intervention in plasma (mmol/L).
Evaluation of liver characteristics profile | 150
  Uric acid, aspartate aminotransferase (ASAT), alanine aminotransferase (ALAT), gamma-glutamyltransferase (GGT) after every intervention and wash-out in plasma (mmol/L).

SECONDARY OUTCOMES:
Evaluation of the stool form | 150 days
  Stool form will be assessed using a validated 7-point scale called Bristol Stool Form Scale pre- and post-dietary intervention.
Evaluation of the defecation frequency | 150
  1. Evacuation frequency 7 days before every blood and microbiome sampling.
  2. Evacuation frequency (number of bowel movements per week) pre- and post-dietary intervention.
Evaluation of the gastrointestinal symptoms | 150
  Frequency and severity of the gastrointestinal symptoms (Constipation, Diarrhea, Bloating, Flatulence, Cramps, Stomach pain). Scale of frequency: Never, Less than 10 times a year, Once a month, Once a week, Every day. Scale of severity: I do not have any gastrointestinal symptoms, Mild (does not disturb), Moderate, Strong (disturbs considerably).

CONTACTS AND LOCATIONS:
Overall Officials: Kaarel Adamberg, PhD, Principal Investigator — Center of Food and Fermentation Technologies
Locations (1):
- Center of Food and Fermentation Technologies, Tallinn, Harju, Estonia

IPD SHARING:
Plan to Share IPD: Yes
Anonymized participant data could be made available for subsequent analysis in the mentioned institution (TFTAK). Data made public will include only aggregates or summaries of the collected data.
Supporting Information: Study Protocol